CLINICAL TRIAL: NCT05041816
Title: Peripheral Nerve Responses to Focal Vibration and Implications in Pain and Mobility for Patients With Diabetic Peripheral Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI resigned and the recruitment had not been started.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13593
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: focal vibration; wearable; nerve conduction study; pain; mobility
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A 6-week, single group, repeated measures with double baselines research design to characterize the changes in sensory and motor nerve performance in DPN, and examine the relations between these changes and changes in pain and mobility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Focal vibration group (Experimental): The Myovolt device used in our previous study will be used for focal vibration delivery during week three to six. Participants will wear Myovolt secured by an elastic band, at a location based on therapist and participants preference. During the four weeks of the FV therapy, participants will be asked to use the Myovolt device for up to 0.5-hour per session (each site 10 minutes per session, with one-minute intersession between sites), once in the morning and once in the evening each day, for five days a week. The dosing paradigm was chosen based on the safety and potential effectiveness of the FV therapy, and our preliminary study.
  Interventions: Device: Focal vibration therapy

INTERVENTIONS:
Device: Focal vibration therapy — Myovolt delivers vibration with a frequency between 60-300 Hz, and acceleration force between 1.8g to 19.1g peak to peak. Myovolt intensity will be set to ~up to 2X the participant's initial Myovolt perception threshold (however, the maximum intensity will be limited to 19.1g which is the maximum intensity the device can deliver). If the stimulation does not feel strong, the participant will be asked to manually increase the intensity until it feels strong but comfortable.

SUMMARY:
The purpose of this study is to characterize the changes in peripheral nerve functions (sensory and motor) in patients with diabetic peripheral neuropathy, and examine the relations between the changes in nerve functions and changes in pain and mobility using focal vibration.

DETAILED DESCRIPTION:
Peripheral nerve impairments are highly prevalent in patients with diabetic peripheral neuropathy (DPN) and are associated with pain and poor mobility. While peripheral sensorimotor nerve function is implicated in neuropathy, the mechanism associated with both pain and mobility is not well understood. Even less understood is the interplay between, and responses to, sensory and motor fibers of the affected peripheral nerve. In our previous study, focal vibration (FV) was effective in reducing pain and improving mobility for only a subgroup of participants with DPN. Because FV stimulates both motor and sensory peripheral nerve fibers, when combined with nerve conduction testing, it offers a unique opportunity to study both the sensory and motor peripheral nerve performance and their contribution to pain and mobility in patients with DPN. We are proposing a single group, repeated measured study to: characterize the changes in sensory and motor peripheral nerve functions; examine the association(s) between these changes and changes in pain and mobility, using FV. If successful, this study will provide us with a better understanding of the role played by sensory and motor nerve impairments in pain and mobility for DPN, and support larger clinical studies to optimize nerve function performance and the FV parameters. We will also explore how changes in the peripheral nerve function associate with severity of DPN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes for at least one year;
* Diabetic peripheral neuropathy as defined by failure to sense the 5.07 (10g) monofilament test in one or more of the six sites tested;
* Age 45-80 years old;
* Able to ambulate independently without assistive devices (e.g., walker or crutches) for 30 feet;
* No evidence of neurological (other than peripheral neuropathy) or orthopedic conditions;
* Able to understand English instructions;
* Have normal or corrected vision.

Exclusion Criteria:

* With other non-diabetic causes of neuropathy by history;
* Symptomatic peripheral vascular disease, joint pain, swelling and/or limited range of motion in the lower extremities that interfere with walking;
* Other systemic or local diseases that could interfere with walking assessment
* Amputation in the lower extremities;
* Clinically diagnosed with dementia greater than mild (screened using Montreal Cognitive Assessment (MOCA) <24)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in CMAP | Change from Baseline CMAP measures every 2 weeks for up to 6 weeks
  The peroneal compound muscle action potential (CMAP)
Changes in NCV | Change from Baseline NCV measures every 2 weeks for up to 6 weeks
  The peroneal motor nerve conduction velocity
Changes in SNAP | Change from Baseline SNAP measures every 2 weeks for up to 6 weeks
  The digital sensory nerve action potentials
Changes in BPI-DPN | Change from Baseline BPI-DPN scores every 2 weeks for up to 6 weeks
  The Brief Pain Inventory Short Form for Diabetic Peripheral Neuropathy
Changes in TUG | Change from Baseline TUG scores every 2 weeks for up to 6 weeks
  Timed Up and Go (TUG) test
Changes in NTSS-6 | Change from Baseline NTSS-6 scores every 2 weeks for up to 6 weeks
  The Neuropathy Total Symptom Score - 6-items (NTSS-6), which quantifies frequency and intensity of aching, burning, prickling and lancinating pain, numbness, and allodynia in patients' feet and legs.
Changes in NSS | Change from Baseline NSS scores every 2 weeks for up to 6 weeks
  The Neuropathy Symptom Score (NSS), which quantifies symptoms of motor, sensory, and autonomic deficits.
Changes in NIS | Change from Baseline NIS scores every 2 weeks for up to 6 weeks
  The Neurologic Impairment Score (NIS), composed of a sensory sub-score (which evaluates sensory perceptions to touch, prickling pain, vibration, joint position, and 1- and 10-g monofilaments in the upper and lower extremities) and a motor sub-score (which evaluates cranial nerves, muscle strength, muscle wasting, and deep tendon reflexes in the upper and lower extremities).

CONTACTS AND LOCATIONS:
Overall Officials: Hongwu Wang, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data might be shared with permission from the funder and PI per request.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the 6 weeks study
Access Criteria: Only de-identified data will be shared with permission from the funder and PI per request

REFERENCES:
- [Background] Rippetoe J, Wang H, James SA, Dionne C, Block B, Beckner M. Improvement of Gait after 4 Weeks of Wearable Focal Muscle Vibration Therapy for Individuals with Diabetic Peripheral Neuropathy. J Clin Med. 2020 Nov 22;9(11):3767. doi: 10.3390/jcm9113767. PMID 33266464
- [Background] Chandrashekhar R, Wang H, Dionne C, James S, Burzycki J. Wearable Focal Muscle Vibration on Pain, Balance, Mobility, and Sensation in Individuals with Diabetic Peripheral Neuropathy: A Pilot Study. Int J Environ Res Public Health. 2021 Mar 2;18(5):2415. doi: 10.3390/ijerph18052415. PMID 33801216